CLINICAL TRIAL: NCT00637533
Title: A Pilot Clinical Trial of Sympathetic Blockade With Botulinum Toxin Type A to Treat Complex Regional Pain Syndrome (CRPS): a Randomized, Double-Blind, Controlled, Crossover Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Ian R Carroll, Stanford University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SU-03102008-1034
Record Dates: First submitted 2008-03-11; First posted 2008-03-18 (Estimated); Last update posted 2011-01-19 (Estimated); Status verified 2011-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Botulinum Toxins, Type A

ARMS (2):
- Placebo (Placebo Comparator): Saline injection
  Interventions: Procedure: Lumbar sympathetic block with Botulinum Toxin type A
- Botulinum Toxin Type A (Experimental): Sympathetic Blockade containing Botulinum Toxin Type A
  Interventions: Procedure: Lumbar sympathetic block with Botulinum Toxin type A

INTERVENTIONS:
Procedure: Lumbar sympathetic block with Botulinum Toxin type A

SUMMARY:
Lumbar sympathetic blocks are part of the standard of care for treating patients with sympathetically-maintained pain (e.g. in complex regional pain syndrome or reflex sympathetic dystrophy- RSD). In these patients lower extremity pain can be reduced or abolished temporarily by blocking sympathetic nerves by doing a lumbar sympathetic block. Patients who respond only transiently to sympathetic blocks often choose between potentially dangerous lumbar sympathetic block with neurolytic agents, surgical sympathectomy, continued severe refractory debilitating pain or other risky invasive surgical procedures such as spinal cord electrical stimulation.. It is hypothesized that Botulinum Toxin Type A (BTA) injected in a lumbar sympathetic block can provide extended sympathetic blockade and thus pain relief. This pilot study aims to see if BTA can be used safely in lower extremity sympathetic blocks, and might be useful in providing prolonged pain relief.

DETAILED DESCRIPTION:
Lumbar sympathetic block will be performed twice on each patient: once as in the standard of practice with 10 cc 0.5% Bupivicaine and once with 75 units of Botox in 10cc of 0.5% Bupivicaine. These will be done in random order and the investigator and the patient will be blinded to which medicine they received. Two weeks after their pain has returned to 75% of their baseline they will receive the second of the blocks.

Lumbar sympathetic blockade in the standard fashion is accomplished by placing an IV in the patient. The patient is then placed face down on a fluoroscopy table. They are then prepped and draped in a sterile fashion. Conscious sedation is provided with versed and Fentanyl in the operating room with monitoring of blood pressure, pulse oximetry, and ekg. The skin is topicalized with one cc of 1% Lidocaine. The L2 lumbar vertebral body is identified and under fluoroscopic guidance a 22 gauge 6 inch spinal needle is placed at the anterolateral border of the L2 vertebral body. The retroperitoneal space is identified with a loss of resistance technique. Correct needle positioned is confirmed radiographically and appropriate spread of medications is verified by injecting 3 cc of radio opaque contrast material. The needle will be aspirated to verify that it is not intravascular. Ten cc of Bupivicaine 0.5% will then be injected in divided dose to ensure safety. Between injections the patient will be asked to report ringing in the ears or tingling in the mouth.

Subjects will be given a form asking them to rate their pain (from 0 to 10 where 0 is no pain and 10 is worst pain imaginable) at noon every day starting one week before the injection and continuing until they feel there pain has returned to baseline or two weeks whichever is longer. Days of analgesia will be the primary endpoint of the study.

ELIGIBILITY:
Inclusion Criteria:Severe pain in a lower extremity (greater than 6/10) of duration more than 6 months despite aggressive previous therapy including both previous lumbar sympathetic block, and previous trial of at least 4 different pain medications including at least 2 of the following: gabapentin, amitryptiline, desipramine, nortryptiline, imipramine, carbamazepine, valproic acid, mexiletine, oxcarbazepine, topiramate, lamotrigine, flecainide, zonisamide, venlafaxine and levetiracetam.

The severity of the pain must be such that the patient must perceive the function of the lower extremity to be compromised by the pain. Exclusion Criteria:Any neuromuscular disorder such as myasthenia gravis, eaton lambert, muscular dystrophy. Any ongoing legal action related to their pain. Any ongoing disability claim. A history of any severe psychiatric disorder. History of any adverse reaction to botulinum toxin. History of botulism. Untreated infection. Coagulopathy. Concurrent use of anticoagulant medications.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2004-05; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Days of Analgesia | Duration of Trial

SECONDARY OUTCOMES:
VAS Pain Score x Time | Duration of trial

CONTACTS AND LOCATIONS:
Overall Officials: Ian R Carroll, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Result] Carroll I, Clark JD, Mackey S. Sympathetic block with botulinum toxin to treat complex regional pain syndrome. Ann Neurol. 2009 Mar;65(3):348-51. doi: 10.1002/ana.21601. PMID 19334078